CLINICAL TRIAL: NCT03356899
Title: Dosage of Intrathecal Hyperbaric Bupivacaine and the Incidence of Post Spinal Shivering in Cesarean Section: is There a Relation?
Brief Title: Dosage of Intrathecal Hyperbaric Bupivacaine and the Incidence of Post Spinal Shivering.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Dr Ezzeldin Ibrahim, Assistant Professor in anaesthesia, intensive care, and pain medicine., Menoufia University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: MenoufiaU2015/2
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Cesarean Section; Shivering
MeSH Terms: interventions — Bupivacaine; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose bupivacaine 0.5% (8mg) (Active Comparator): Bupivacaine 0.5% for spinal anesthesia
  Interventions: Drug: Low dose bupivacaine 0.5% (8mg)
- High dose bupivacaine 0.5% (10mg) (Active Comparator): Bupivacaine 0.5% for spinal anesthesia
  Interventions: Drug: High dose bupivacaine 0.5% (10mg)

INTERVENTIONS:
Drug: Low dose bupivacaine 0.5% (8mg) — 8 mg hyperbaric bupivacaine with added 25 µg fentanyl to form a total volume of 2.1 ml
  Other Names: Bupivacaine for spinal anaesthesia.
  Arms: Low dose bupivacaine 0.5% (8mg)
Drug: High dose bupivacaine 0.5% (10mg) — 10 mg hyperbaric bupivacaine with added 25 µg fentanyl to form a total volume of 2.5
  Other Names: Bupivacaine for spinal anaesthesia
  Arms: High dose bupivacaine 0.5% (10mg)

SUMMARY:
Shivering is very common after spinal anaesthesia. Many studies have investigated the role of adding adjuvants to the local anaesthetics to decrease the incidence of post-spinal shivering. Non of the studies n the literature review have investigated the role of different dose of local anaesthetic alone in reducing the incidence of post-spinal shivering. In the present study the investigators aimed to compare the effect of different local anaesthetic dose in reducing post-spinal shivering.

DETAILED DESCRIPTION:
After approval of the ethics committee, department of anaesthesia, Menoufia University and written informed consent, a hundred full-term pregnant ladies undergoing elective cesarean section were enrolled in this study.

The pregnant ladies were randomly assigned using a computerised software to one of two groups, low dose bupivacaine (LB) and high dose bupivacaine (HB), 50 patients each according to bupivacaine dose. Group LB received low dose bupivacaine (8 mg hyperbaric bupivacaine) Group HB received high dose bupivacaine (10 mg hyperbaric bupivacaine).

Vital signs including heart rate and mean arterial blood pressure intra-operatively until the end of surgery.

The severity of shivering was the primary endpoint. Shivering was graded using a scale: 0, no shivering; 1, piloerection but no visible muscle activity; 2, muscular activity in one group of muscle; 3, muscular activity in more than one muscle group but not generalized movement; and 4, shivering involving the movement of the whole body. Shivering score was recorded for the whole study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 22 and 35 year old, and American Society of Anesthetists (ASA) I or II were included in the study and consented to have spinal anaesthesia for their section.

Exclusion Criteria:

* Patients who had contraindication to spinal anesthesia, high-risk pregnancy, history of seizures, mental illness, acute fetal distress, and patients refused spinal anesthesia were excluded from the study.

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All patients were females scheduled for elective caesarian section.
Enrollment: 100 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-09-29 (Actual)

PRIMARY OUTCOMES:
Shivering score | Peri-operatively
  Shivering score is a graded score using a scale: 0, no shivering; 1, piloerection but no visible muscle activity; 2, muscular activity in one group of muscle; 3, muscular activity in more than one muscle group but not generalised movement; and 4, shivering involving the movement of the whole body.

SECONDARY OUTCOMES:
Mean arterial blood pressure (mmHg) | Peri-operatively
  Mean arterial blood pressure reading
Heart rate (beat/minute) | Peri-operatively
  The number of hear beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Ezzeldin Ibrahim, PhD, Principal Investigator — Professor
Locations (1):
- Faculty of Medicine, Menoufia Univeristy, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No